CLINICAL TRIAL: NCT04662008
Title: CLOSER_MS: Communicating With Local or Distance Caregivers Offering Support and Electronic Resources
Brief Title: Offering Support and Electronic Resources for Care Partners of Those With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MS-1610-37015 enhancement
Record Dates: First submitted 2020-12-02; First posted 2020-12-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis; Caregivers
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High resource tailored intervention (Active Comparator): Tele-coaching arm
  Interventions: Behavioral: Tele-coaching; Behavioral: Website
- Low-resource web-only intervention (Active Comparator): Website arm
  Interventions: Behavioral: Website

INTERVENTIONS:
Behavioral: Tele-coaching — This intervention arm will receive 4 one-to-one tele-coaching sessions facilitated by an advanced practice social worker. The sessions will take place over a 6-week period and will begin with a needs assessments to allow for tailoring of the intervention sessions. The sessions will include information and support in the areas of: general MS information, strategies for caring for a loved one with MS, MS and Covid (care strategies), caring for yourself, and planning for the future. The intervention will take place using Zoom videoconferencing technology or via telephone- per subject preference. In addition, all subjects will receive access to a study-specific website. The website will have links to publicly available information including general information about MS, online information, self-care, communication, caregiving, COVID-19, future planning.
  Arms: High resource tailored intervention
Behavioral: Website — This intervention arm will receive access to a study-specific website. The website will have links to publicly available information including: general information about MS, online information, self-care, communication, caregiving, COVID-19, future planning.

SUMMARY:
This study is an enhancement of the Fatigue Management Programs for People with MS study (NCT03550170). The purpose of this randomized clinical trial is to test the effectiveness of two interventions delivered remotely to support unpaid caregivers (UC) of people with multiple sclerosis (MS). We hypothesize that a high resource intervention will be significantly better than a lower resource intervention in terms of the primary outcome (UC anxiety, depression, and stress) and secondary outcome (COVID specific anxiety).

DETAILED DESCRIPTION:
UCs are often caring for persons with chronic disabling conditions, who are at higher risk for severe COVID-19 illness. This presents incredibly stressful situations for UCs, which can result in depression, anxiety, and worse health outcomes both for them and their care recipients. Until a vaccine becomes available, these demands will force UCs to provide more support, whether in-person or remotely, for persons with MS. The aim of this study is to compare 2 modes of supporting UCs of people with MS. We will compare the effectiveness of a high resource highly tailored intervention that includes tele-coaching intervention (delivered via videoconference or phone) + web site information to a low-resource web-site only intervention. Our primary outcomes are UC anxiety, depression, and stress (DASS-42 scale) and a secondary outcome is COVID specific anxiety (CAS scale). These 2 interventions were selected because they will inform administrators and clinicians on whether a resource-intensive or a low-resource intervention is needed to yield meaningful outcomes. The comparison will also help UC decide how they should spend their limited time. These interventions are relevant to UCs of people with MS because of their need for tailored information provided in flexible ways to promote learning and support.

ELIGIBILITY:
Inclusion Criteria:

1. An adult family member or friend (18 years of age or older) of a person with MS
2. Self-identified as an unpaid caregiver for person with MS
3. Access to internet
4. Capable of providing informed consent in English

Exclusion Criteria:

1. Under age 18
2. Cannot speak English
3. Unable to provide consent
4. No access to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
anxiety, depression, and stress (DASS-42) | Each subject will be given the assessments at 3 points during the study: baseline, 6 weeks, and 12 weeks
  Change from baseline in anxiety, depression, and stress levels. Each of the three DASS scales contains 14 items. Using a 4-point Likert scale, scores range from 0- 42 for each scale. Higher scores indicate more depression, anxiety, and stress.

SECONDARY OUTCOMES:
COVID specific anxiety (CAS scale) | Each subject will be given the assessments at 3 points during the study: baseline, 6 weeks, and 12 weeks
  Change from baseline in COVID specific anxiety. Using a 5-point scale, from 0 (not at all) to 4 (nearly every day), total score ranges from 0-20 while individual items range from 0-4. Higher scores indicate higher anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Douglas SL, Plow M, Packer T, Lipson AR, Lehman MJ. Psychoeducational Interventions for Caregivers of Persons With Multiple Sclerosis: Protocol for a Randomized Trial. JMIR Res Protoc. 2021 Aug 26;10(8):e30617. doi: 10.2196/30617. PMID 34435971